CLINICAL TRIAL: NCT01717391
Title: Improving Pelvic Cancer Patient Chemoradiotherapy Outcomes With FLT PET Imaging
Brief Title: [F-18] Fluorothymidine PET/CT Imaging for Pelvic Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John M. Buatti (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, John M. Buatti, Professor of Radiation Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201204712; R01CA169336 (NIH)
Record Dates: First submitted 2012-10-18; First posted 2012-10-30 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Uterine Cervical Neoplasms; Endometrial Neoplasms; Anus Neoplasms; Rectal Neoplasms; Prostatic Neoplasms
Keywords: radiotherapy; Positron-Emission Tomography and Computed Tomography; chemotherapy; bone marrow
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Anus Neoplasms; Rectal Neoplasms; Prostatic Neoplasms | interventions — alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fluorothymidine F 18 PET/CT (Experimental): Fluorothymidine F 18 (FLT) PET/CT imaging ordered pre-radiation therapy, during weeks 1 and 2 of radiation therapy, and then at 1 month and 12 months after radiation therapy. The FLT PET/CT imaging ordered pre-radiation therapy is used for bone marrow sparing IMRT radiation therapy.
  Interventions: Drug: fluorothymidine F 18

INTERVENTIONS:
Drug: fluorothymidine F 18 — A patient-specific bone marrow map will be designed from the pre-therapy FLT PET/CT imaging. A highly conformal radiation plan will be designed to spare active bone marrow.
  Other Names: [F-18] Fluorothymidine

SUMMARY:
[F-18] Fluorothymidine PET imaging will be used to create a radiation therapy treatment plan to avoid active bone marrow in the pelvis. This will be done to evaluate if sparing bone marrow will help maintain blood counts. This would impact chemotherapy administration.

DETAILED DESCRIPTION:
Overall survival of pelvic cancer patients depends on control of systemic disease. If local radiation therapy depletes bone marrow function to such an extent that systemic therapies must be withheld, chances of metastatic failure increase significantly. This may be more significant for this group of patients because approximately one third of adult bone marrow is located in the pelvic region. Strategies to minimize toxicities would benefit a range of pelvic cancer patients including gynecologic, anal, rectal, and prostate. New chemoradiation combinations improve outcomes for these disease sites, but come at the cost of higher levels of toxicity. As many as 40% of cervical cancer patients miss at least one chemotherapy cycle due to hematologic toxicity and 36% of anal cancer patients experience grade 3 or 4 hematologic toxicity when undergoing chemoradiation therapy. A clinical trial of concurrent chemoradiation therapy for rectal cancer was terminated due to toxicity, including hematologic toxicities. Concurrent chemoradiation therapy shows promise for advanced stage prostate cancers, but it also increases grade 3 and 4 toxicities. To successfully limit hematologic toxicities for pelvic cancers, it is extremely advantageous to avoid irradiating the highly proliferative compartments of the pelvic bone marrow. However, the complex structure of the pelvis makes it difficult to assess the efficacy of radiation therapy (RT) planning strategies to avoid areas critical to hematopoiesis. Uptake of [18F]fluorothymidine imaged with positron emission tomography (FLT PET/CT) can be an accurate and sensitive tool for identifying and monitoring the effects of chemoradiation on proliferative pelvic bone marrow. Clinically validating the utility of FLT PET/CT imaging for identifying active bone marrow in the design of bone marrow sparing RT-plans and the important bone marrow assessment time points would provide a method to reduce acute and chronic hematologic toxicities for pelvic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Recommended to undergo pelvic irradiation with concurrent chemotherapy.
* At least 18 years of age. Pediatrics would be best served by a protocol designed for their specific needs.
* Karnofsky Performance Status of at least 60% at time of screening.
* Life expectancy of greater than 6 months.
* Subject must have normal organ and marrow function (as defined below) within 30 days of study enrollment:

  * leukocytes at least 3,000 / µL
  * absolute neutrophil count of at least 1500 / µL
  * platelets of at least 100,000 / µL
  * creatinine equal to or less than the upper limit of normal
* not pregnant (as applicable)

Exclusion Criteria:

* history of allergic reactions attributed to compounds of similar chemical or biologic composition to FLT
* an oncology research protocol requiring full pelvic radiation (i.e., 4 field box technique)
* uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* subjects taking nucleoside analog medications such as those used as antiretroviral agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10-01; Primary Completion 2016-02-29 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Buatti, PhD, Principal Investigator — Department of Radiation Oncology, The University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon request. A contract may need to be put into place, dependent upon data shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Email the principal investigator for access.

REFERENCES:
- [Background] McGuire SM, Menda Y, Ponto LL, Gross B, Juweid M, Bayouth JE. A methodology for incorporating functional bone marrow sparing in IMRT planning for pelvic radiation therapy. Radiother Oncol. 2011 Apr;99(1):49-54. doi: 10.1016/j.radonc.2011.01.025. Epub 2011 Mar 22. PMID 21397965
- [Background] McGuire SM, Menda Y, Boles Ponto LL, Gross B, Buatti J, Bayouth JE. 3'-deoxy-3'-[(1)(8)F]fluorothymidine PET quantification of bone marrow response to radiation dose. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):888-93. doi: 10.1016/j.ijrobp.2010.12.009. Epub 2011 Feb 6. PMID 21300484
- [Background] Menda Y, Ponto LL, Dornfeld KJ, Tewson TJ, Watkins GL, Gupta AK, Anderson C, McGuire S, Schultz MK, Sunderland JJ, Graham MM, Buatti JM. Investigation of the pharmacokinetics of 3'-deoxy-3'-[18F]fluorothymidine uptake in the bone marrow before and early after initiation of chemoradiation therapy in head and neck cancer. Nucl Med Biol. 2010 May;37(4):433-8. doi: 10.1016/j.nucmedbio.2010.02.005. PMID 20447554
- [Result] McGuire SM, Bhatia SK, Sun W, Jacobson GM, Menda Y, Ponto LL, Smith BJ, Gross BA, Bayouth JE, Sunderland JJ, Graham MM, Buatti JM. Using [(18)F]Fluorothymidine Imaged With Positron Emission Tomography to Quantify and Reduce Hematologic Toxicity Due to Chemoradiation Therapy for Pelvic Cancer Patients. Int J Radiat Oncol Biol Phys. 2016 Sep 1;96(1):228-39. doi: 10.1016/j.ijrobp.2016.04.009. Epub 2016 Apr 19. PMID 27319286
- [Result] McGuire SM, Menda Y, Ponto LLB, Gross B, TenNapel M, Smith BJ, Bayouth JE. Spatial mapping of functional pelvic bone marrow using FLT PET. J Appl Clin Med Phys. 2014 Jul 8;15(4):129-136. doi: 10.1120/jacmp.v15i4.4780. PMID 25207403

RESULTS

PARTICIPANT FLOW:
Groups:
- FLT PET/CT: FLT PET/CT imaging ordered pre-radiation therapy, during weeks 1 and 2 of radiation therapy, and then at 1 month and 12 months after radiation therapy. The FLT PET/CT imaging ordered pre-radiation therapy is used for bone marrow sparing IMRT radiation therapy.
  Fluorothymidine F 18: A patient-specific bone marrow map will be designed from the pre-therapy FLT PET/CT imaging. A highly conformal radiation plan will be designed to spare active bone marrow.
Period: Overall Study
Arm/Group | FLT PET/CT
Started | 36
Completed | 27
Not Completed | 9
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1
Not completed — FLT technical failure | 3

BASELINE CHARACTERISTICS:
Arm/Group | FLT PET/CT
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Percent Difference From Baseline IMRT Plan (%)
Description: The difference in volume of bone marrow receiving radiation using a bone-marrow-sparing radiation plan compared to a standard radiation plan (IMRT), expressed as a percentage. Both plans are patient-specific. Bone-marrow is identified using the baseline FLT PET/CT obtained pre-imaging. Active bone marrow is considered to have an uptake value (SUV) of 2, 3, or 4. The standard IMRT plan was created using the criteria of the National Cancer Institute's Radiation Therapy Oncology Group study RTOG-0418. Radiation doses evaluated are 5 Gray, 10 Gray, 20 Gray, and 30 Gray. The change in dose to tumor is also provided. A negative value indicates that more bone marrow or tissue was spared using the bone-marrow sparing plan.
Time Frame: Baseline (pre-treatment)
Population: All participants who received an FLT PET/CT during radiation simulation.
Measure: Mean (Standard Deviation); unit: Percent difference (%)
Groups:
- Basline FLT PET/CT (All Subjects): FLT PET/CT imaging ordered pre-radiation therapy to create a patient-specific bone marrow map to spare active bone marrow.
Arm/Group | Basline FLT PET/CT (All Subjects)
Number analyzed (Participants) | 27
Percent difference (%)
  % difference, volume receiving 5 Gray | -4.7 (3.3)
  % difference, volume receiving 10 Gray | -9.3 (4.2)
  % difference, volume receiving 20 Gray | -14.2 (4.1)
  % difference, volume receiving 30 Gray | -13.4 (7.6)
  % difference, dose to target (tumor) volume | -0.1 (0.4)

2. Secondary Outcome: Chemotherapy Compliance
Description: The number of participants who had chemotherapy withheld at least once for low blood counts.
Time Frame: At 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | FLT PET/CT
Number analyzed (Participants) | 27
Participants | 7

3. Secondary Outcome: Number of Participants With Standardized Toxicity Severity Grades for White Blood Cell Counts
Description: White blood cell counts measurements expressed in standardized toxicity severity grades (Common Terminology Criteria for Adverse Events, v4.03) measured weekly during combined chemotherapy and radiation therapy treatment and then once at 30 day follow-up and at 1 year follow-up
Time Frame: baseline, weekly during radiation treatment for up to 5 weeks, 30 days and 1 year after treatment
Population: This group includes all tumor types treated in this clinical trial and provides an overall averages.
Measure: Count of Participants; unit: Participants
Groups:
- Bone-marrow Sparing Radiation Therapy (IMRT): Participants who have undergone the FLT PET/CT imaging ordered pre-radiation therapy to create a patient-specific bone marrow map to spare active bone marrow.
Arm/Group | Bone-marrow Sparing Radiation Therapy (IMRT)
Number analyzed (Participants) | 27
Participants
  Baseline (pre-treatment): Grade 0 (no toxicity) | 27
  Baseline (pre-treatment): CTCAE grade 1 | 0
  Baseline (pre-treatment): CTCAE grade 2 | 0
  Baseline (pre-treatment): CTCAE grade 3 | 0
  Baseline (pre-treatment): CTCAE grade 4 (most severe) | 0
  Baseline (pre-treatment): Not assessed (test omitted) | 0
  Therapy, week 1: Grade 0 (no toxicity) | 27
  Therapy, week 1: CTCAE grade 1 | 0
  Therapy, week 1: CTCAE grade 2 | 0
  Therapy, week 1: CTCAE grade 3 | 0
  Therapy, week 1: CTCAE grade 4 (most severe) | 0
  Therapy, week 1: Not assessed (test omitted) | 0
  Therapy, week 2: Grade 0 (no toxicity) | 15
  Therapy, week 2: CTCAE grade 1 | 7
  Therapy, week 2: CTCAE grade 2 | 1
  Therapy, week 2: CTCAE grade 3 | 3
  Therapy, week 2: CTCAE grade 4 (most severe) | 1
  Therapy, week 2: Not assessed (test omitted) | 0
  Therapy, week 3: Grade 0 (no toxicity) | 13
  Therapy, week 3: CTCAE grade 1 | 5
  Therapy, week 3: CTCAE grade 2 | 2
  Therapy, week 3: CTCAE grade 3 | 1
  Therapy, week 3: CTCAE grade 4 (most severe) | 0
  Therapy, week 3: Not assessed (test omitted) | 6
  Therapy, week 4: Grade 0 (no toxicity) | 13
  Therapy, week 4: CTCAE grade 1 | 5
  Therapy, week 4: CTCAE grade 2 | 4
  Therapy, week 4: CTCAE grade 3 | 2
  Therapy, week 4: CTCAE grade 4 (most severe) | 0
  Therapy, week 4: Not assessed (test omitted) | 3
  Therapy, week 5: Grade 0 (no toxicity) | 10
  Therapy, week 5: CTCAE grade 1 | 3
  Therapy, week 5: CTCAE grade 2 | 3
  Therapy, week 5: CTCAE grade 3 | 1
  Therapy, week 5: CTCAE grade 4 (most severe) | 0
  Therapy, week 5: Not assessed (test omitted) | 10
  30 days post-therapy: Grade 0 (no toxicity) | 20
  30 days post-therapy: CTCAE grade 1 | 2
  30 days post-therapy: CTCAE grade 2 | 0
  30 days post-therapy: CTCAE grade 3 | 0
  30 days post-therapy: CTCAE grade 4 (most severe) | 0
  30 days post-therapy: Not assessed (test omitted) | 5
  1 year post-therapy: Grade 0 (no toxicity) | 16
  1 year post-therapy: CTCAE grade 1 | 1
  1 year post-therapy: CTCAE grade 2 | 1
  1 year post-therapy: CTCAE grade 3 | 0
  1 year post-therapy: CTCAE grade 4 (most severe) | 0
  1 year post-therapy: Not assessed (test omitted) | 9

4. Secondary Outcome: Number of Participants With Standardized Toxicity Severity Grades for Decreased Platelet Counts.
Description: Platelet cell counts measurements expressed in standardized toxicity severity grades (Common Terminology Criteria for Adverse Events, v4.03) measured once weekly during combined chemotherapy and radiation therapy, then once at 30 day follow-up, and once at 1 year follow-up
Time Frame: baseline, weekly during radiation treatment for up to 5 weeks, 30 days and 1 year after treatment
Population: This group includes all tumor types treated in this clinical trial and provides an overall averages.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-marrow Sparing Radiation Therapy (IMRT)
Number analyzed (Participants) | 27
Participants
  Baseline (pre-treatment): CTCAE grade 0 (no toxicity) | 27
  Baseline (pre-treatment): CTCAE grade 1 | 0
  Baseline (pre-treatment): CTCAE grade 2 | 0
  Baseline (pre-treatment): CTCAE grade 3 | 0
  Baseline (pre-treatment): CTCAE grade 4 (severe toxicity) | 0
  Baseline (pre-treatment): Not assessed (test omitted) | 0
  Therapy, week 1: CTCAE grade 0 (no toxicity) | 27
  Therapy, week 1: CTCAE grade 1 | 0
  Therapy, week 1: CTCAE grade 2 | 0
  Therapy, week 1: CTCAE grade 3 | 0
  Therapy, week 1: CTCAE grade 4 (severe toxicity) | 0
  Therapy, week 1: Not assessed (test omitted) | 0
  Therapy, week 2: CTCAE grade 0 (no toxicity) | 16
  Therapy, week 2: CTCAE grade 1 | 9
  Therapy, week 2: CTCAE grade 2 | 0
  Therapy, week 2: CTCAE grade 3 | 2
  Therapy, week 2: CTCAE grade 4 (severe toxicity) | 0
  Therapy, week 2: Not assessed (test omitted) | 0
  Therapy, week 3: CTCAE grade 0 (no toxicity) | 12
  Therapy, week 3: CTCAE grade 1 | 6
  Therapy, week 3: CTCAE grade 2 | 1
  Therapy, week 3: CTCAE grade 3 | 1
  Therapy, week 3: CTCAE grade 4 (severe toxicity) | 0
  Therapy, week 3: Not assessed (test omitted) | 7
  Therapy, week 4: CTCAE grade 0 (no toxicity) | 15
  Therapy, week 4: CTCAE grade 1 | 6
  Therapy, week 4: CTCAE grade 2 | 2
  Therapy, week 4: CTCAE grade 3 | 0
  Therapy, week 4: CTCAE grade 4 (severe toxicity) | 0
  Therapy, week 4: Not assessed (test omitted) | 4
  Therapy, week 5: CTCAE grade 0 (no toxicity) | 9
  Therapy, week 5: CTCAE grade 1 | 7
  Therapy, week 5: CTCAE grade 2 | 1
  Therapy, week 5: CTCAE grade 3 | 0
  Therapy, week 5: CTCAE grade 4 (severe toxicity) | 0
  Therapy, week 5: Not assessed (test omitted) | 10
  30 days post-therapy: CTCAE grade 0 (no toxicity) | 17
  30 days post-therapy: CTCAE grade 1 | 4
  30 days post-therapy: CTCAE grade 2 | 1
  30 days post-therapy: CTCAE grade 3 | 0
  30 days post-therapy: CTCAE grade 4 (severe toxicity) | 0
  30 days post-therapy: Not assessed (test omitted) | 5
  1 year post-therapy: CTCAE grade 0 (no toxicity) | 16
  1 year post-therapy: CTCAE grade 1 | 2
  1 year post-therapy: CTCAE grade 2 | 0
  1 year post-therapy: CTCAE grade 3 | 0
  1 year post-therapy: CTCAE grade 4 (severe toxicity) | 0
  1 year post-therapy: Not assessed (test omitted) | 9

5. Secondary Outcome: Number of Participants With Standardized Toxicity Severity Grades for Decreased Absolute Neutrophil Counts (ANCs)
Description: Absolute neutrophil counts (ANCs) measurements expressed in standardized toxicity severity grades (Common Terminology Criteria for Adverse Events, v4.03) measured once weekly during combined chemotherapy and radiation therapy, then once at 30 day follow-up, and once at 1 year follow-up
Time Frame: baseline, weekly during radiation treatment for up to 5 weeks, 30 days and 1 year after treatment
Population: This group includes all tumor types treated in this clinical trial and provides an overall averages.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-marrow Sparing Radiation Therapy (IMRT)
Number analyzed (Participants) | 27
Participants
  Baseline (pre-treatment): CTCAE grade 0 (no toxicity) | 27
  Baseline (pre-treatment): CTCAE grade 1 | 0
  Baseline (pre-treatment): CTCAE grade 2 | 0
  Baseline (pre-treatment): CTCAE grade 3 | 0
  Baseline (pre-treatment): CTCAE grade 4 (most severe) | 0
  Baseline (pre-treatment): Not assessed (test omitted) | 0
  Therapy, week 1: CTCAE grade 0 (no toxicity) | 25
  Therapy, week 1: CTCAE grade 1 | 2
  Therapy, week 1: CTCAE grade 2 | 0
  Therapy, week 1: CTCAE grade 3 | 0
  Therapy, week 1: CTCAE grade 4 (most severe) | 0
  Therapy, week 1: Not assessed (test omitted) | 0
  Therapy, week 2: CTCAE grade 0 (no toxicity) | 16
  Therapy, week 2: CTCAE grade 1 | 8
  Therapy, week 2: CTCAE grade 2 | 0
  Therapy, week 2: CTCAE grade 3 | 1
  Therapy, week 2: CTCAE grade 4 (most severe) | 2
  Therapy, week 2: Not assessed (test omitted) | 0
  Therapy, week 3: CTCAE grade 0 (no toxicity) | 16
  Therapy, week 3: CTCAE grade 1 | 4
  Therapy, week 3: CTCAE grade 2 | 0
  Therapy, week 3: CTCAE grade 3 | 1
  Therapy, week 3: CTCAE grade 4 (most severe) | 0
  Therapy, week 3: Not assessed (test omitted) | 6
  Therapy, week 4: CTCAE grade 0 (no toxicity) | 17
  Therapy, week 4: CTCAE grade 1 | 5
  Therapy, week 4: CTCAE grade 2 | 2
  Therapy, week 4: CTCAE grade 3 | 0
  Therapy, week 4: CTCAE grade 4 (most severe) | 0
  Therapy, week 4: Not assessed (test omitted) | 3
  Therapy, week 5: CTCAE grade 0 (no toxicity) | 13
  Therapy, week 5: CTCAE grade 1 | 2
  Therapy, week 5: CTCAE grade 2 | 2
  Therapy, week 5: CTCAE grade 3 | 0
  Therapy, week 5: CTCAE grade 4 (most severe) | 0
  Therapy, week 5: Not assessed (test omitted) | 10
  30 days post-therapy: CTCAE grade 0 (no toxicity) | 21
  30 days post-therapy: CTCAE grade 1 | 1
  30 days post-therapy: CTCAE grade 2 | 0
  30 days post-therapy: CTCAE grade 3 | 0
  30 days post-therapy: CTCAE grade 4 (most severe) | 0
  30 days post-therapy: Not assessed (test omitted) | 5
  1 year post-therapy: CTCAE grade 0 (no toxicity) | 16
  1 year post-therapy: CTCAE grade 1 | 2
  1 year post-therapy: CTCAE grade 2 | 0
  1 year post-therapy: CTCAE grade 3 | 0
  1 year post-therapy: CTCAE grade 4 (most severe) | 0
  1 year post-therapy: Not assessed (test omitted) | 9

6. Secondary Outcome: Number of Participants With Standardized Toxicity Severity Grades for Decreased Lymphocyte Counts.
Description: Lymphocyte counts measurements expressed in standardized toxicity severity grades (Common Terminology Criteria for Adverse Events, v4.03) measured once weekly during combined chemotherapy and radiation therapy, then once at 30 day follow-up, and once at 1 year follow-up
Time Frame: baseline, weekly during radiation treatment for up to 5 weeks, 30 days and 1 year after treatment
Population: This group includes all tumor types treated in this clinical trial and provides an overall averages.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-marrow Sparing Radiation Therapy (IMRT)
Number analyzed (Participants) | 27
Participants
  Baseline (pre-treatment): CTCAE grade 0 (no toxicity) | 27
  Baseline (pre-treatment): CTCAE grade 1 | 0
  Baseline (pre-treatment): CTCAE grade 2 | 0
  Baseline (pre-treatment): CTCAE grade 3 | 0
  Baseline (pre-treatment): CTCAE grade 4 (most severe) | 0
  Baseline (pre-treatment): Not assessed (test omitted) | 0
  Therapy, week 1: CTCAE grade 0 (no toxicity) | 25
  Therapy, week 1: CTCAE grade 1 | 2
  Therapy, week 1: CTCAE grade 2 | 0
  Therapy, week 1: CTCAE grade 3 | 0
  Therapy, week 1: CTCAE grade 4 (most severe) | 0
  Therapy, week 1: Not assessed (test omitted) | 0
  Therapy, week 2: CTCAE grade 0 (no toxicity) | 16
  Therapy, week 2: CTCAE grade 1 | 8
  Therapy, week 2: CTCAE grade 2 | 0
  Therapy, week 2: CTCAE grade 3 | 1
  Therapy, week 2: CTCAE grade 4 (most severe) | 2
  Therapy, week 2: Not assessed (test omitted) | 0
  Therapy, week 3: CTCAE grade 0 (no toxicity) | 16
  Therapy, week 3: CTCAE grade 1 | 4
  Therapy, week 3: CTCAE grade 2 | 0
  Therapy, week 3: CTCAE grade 3 | 1
  Therapy, week 3: CTCAE grade 4 (most severe) | 0
  Therapy, week 3: Not assessed (test omitted) | 6
  Therapy, week 4: CTCAE grade 0 (no toxicity) | 17
  Therapy, week 4: CTCAE grade 1 | 5
  Therapy, week 4: CTCAE grade 2 | 2
  Therapy, week 4: CTCAE grade 3 | 0
  Therapy, week 4: CTCAE grade 4 (most severe) | 0
  Therapy, week 4: Not assessed (test omitted) | 3
  Therapy, week 5: CTCAE grade 0 (no toxicity) | 13
  Therapy, week 5: CTCAE grade 1 | 2
  Therapy, week 5: CTCAE grade 2 | 2
  Therapy, week 5: CTCAE grade 3 | 0
  Therapy, week 5: CTCAE grade 4 (most severe) | 0
  Therapy, week 5: Not assessed (test omitted) | 10
  30 days post-therapy: CTCAE grade 0 (no toxicity) | 21
  30 days post-therapy: CTCAE grade 1 | 1
  30 days post-therapy: CTCAE grade 2 | 0
  30 days post-therapy: CTCAE grade 3 | 0
  30 days post-therapy: CTCAE grade 4 (most severe) | 0
  30 days post-therapy: Not assessed (test omitted) | 5
  1 year post-therapy: CTCAE grade 0 (no toxicity) | 16
  1 year post-therapy: CTCAE grade 1 | 2
  1 year post-therapy: CTCAE grade 2 | 0
  1 year post-therapy: CTCAE grade 3 | 0
  1 year post-therapy: CTCAE grade 4 (most severe) | 0
  1 year post-therapy: Not assessed (test omitted) | 9

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 48 hours after injection with FLT, the investigational drug under study.
Description: Adverse events were collected through medical chart review as well as by direct contact by a licensed health provider with participant for their perceived side effects from the FLT PET/CT scan. Chart review is considered non-systematic collection; the semi-structured interview 48 hours after the scan is considered a systematic collection. Grade 0 is considered no toxicity (symptom is absent) and grade 4 is considered the most severe toxicity.
Arm/Group | FLT PET/CT
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 6/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLT PET/CT (N=27)
Diarrhea, grade 1 (Gastrointestinal disorders) | 3 (5)
Diarrhea, grade 2 (Gastrointestinal disorders) | 2 (2)
Nausea, grade 1 (Gastrointestinal disorders) | 6 (6)
Headache, grade 1 (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes